CLINICAL TRIAL: NCT03583450
Title: Perioperative Virtual Reality for Pediatric Anesthesia: Pediatric Distraction on Induction With Virtual Reality (PEDI-VR)
Brief Title: Perioperative Virtual Reality for Pediatric Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-25277
Record Dates: First submitted 2018-06-18; First posted 2018-07-11 (Actual); Results first posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Anxiety
Keywords: Virtual Reality; Pediatric Anesthesia
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Perioperative virtual reality headset (Experimental): Perioperative virtual reality headset with mobile app and routine anesthetic care
  Interventions: Device: Perioperative virtual reality headset with mobile app
- Control (No Intervention): Routine anesthetic care

INTERVENTIONS:
Device: Perioperative virtual reality headset with mobile app — Perioperative virtual reality headset with mobile app (Samsung Gear VR headset, ChariotVR software)
  Arms: Perioperative virtual reality headset

SUMMARY:
The goal of this study is to evaluate the use of immersive audiovisual distraction and virtual reality to reduce perioperative anxiety in pediatric patients undergoing surgery at UCSF Benioff Children's Hospital. The study plans to employ virtual reality headsets during induction of anesthesia in pediatric patients for elective surgery in a randomized clinical trial.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the use of immersive audiovisual distraction and virtual reality to reduce perioperative anxiety in pediatric patients undergoing surgery at UCSF Benioff Children's Hospital. The study plans to employ virtual reality headsets during induction of anesthesia in pediatric patients for elective surgery in a randomized clinical trial. We will be enrolling patients age 5-12 years presenting for elective surgery.

Patients will be randomized to one of two groups: (1) virtual reality headset with routine anesthetic care and (2) routine anesthetic care only.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 5-12 years
* Patients present in preoperative area for induction of general anesthesia for an elective surgery or procedure

Exclusion Criteria:

* Patients with injuries to the head/face that would prohibit wearing of headsets
* Patients with loss of consciousness, altered mental status, life-threatening injuries/illness or multi-trauma
* Patients with open skin, lice, scabies, or other infectious skin conditions on the head/face
* Patients with a history of or current symptoms of vertigo
* Patients who are blind
* Patients with significant developmental or cognitive delays who may not be able to engage with or tolerate the virtual reality environment, as determined by their parent/caregiver
* Patients on whom the VR headset does not fit appropriately
* Non-English speaking patients (due to limited availability of non-English study documents and consents)

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Jung, Principal Investigator — UCSF Medical Center; Jina Sinskey, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Benioff Children's Hospital, San Francisco, California, United States

REFERENCES:
- [Derived] Jung MJ, Libaw JS, Ma K, Whitlock EL, Feiner JR, Sinskey JL. Pediatric Distraction on Induction of Anesthesia With Virtual Reality and Perioperative Anxiolysis: A Randomized Controlled Trial. Anesth Analg. 2021 Mar 1;132(3):798-806. doi: 10.1213/ANE.0000000000005004. PMID 32618627

RESULTS

PARTICIPANT FLOW:
Groups:
- Perioperative Virtual Reality Headset: Perioperative virtual reality headset with mobile app (Samsung Gear VR headset, ChariotVR software) with routine anesthetic care
Period: Overall Study
Arm/Group | Perioperative Virtual Reality Headset | Control
Started | 34 | 37
Completed | 33 | 37
Not Completed | 1 | 0
Not completed — hardware malfunction (battery depletion) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perioperative Virtual Reality Headset | Control | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (2.3) | 7.8 (2.3) | 8.0 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 16 | 19 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 5 | 3 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 20 | 19 | 39
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 6 | 11 | 17
Region of Enrollment [Number; unit: participants]
  United States | 34 | 37 | 71
Height [Mean (Standard Deviation); unit: cm] | 131.8 (12.8) | 130.2 (15.5) | 131.0 (14.2)
Weight [Mean (Standard Deviation); unit: kg] | 32.9 (11.9) | 31.9 (15.2) | 32.4 (13.6)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 18.5 (4.0) | 18.0 (4.8) | 18.2 (4.4)
ASA physical status classification [Count of Participants; unit: Participants] — The ASA Physical Status Classification System is used to assess and communicate a patient's pre-anesthesia medical co-morbidities. ASA I is the healthiest and ASA VI is a declared brain-dead patient.
  * ASA I: Normal healthy patient
  * ASA II: Patient with mild systemic disease
  * ASA III: Patient with severe systemic disease
  Participants
    ASA 1 | 11 | 15 | 26
    ASA 2 | 16 | 18 | 34
    ASA 3 | 7 | 4 | 11
Prior general anesthesia [Count of Participants; unit: Participants]
  Yes | 19 | 18 | 37
  No | 15 | 19 | 34
Number of prior general anesthetics [Mean (Standard Deviation); unit: Prior general anesthetics] | 3.3 (4.1) | 2.7 (5.2) | 3.0 (4.7)
Modified Yale Preoperative Anxiety Scale in preop [Median (Inter-Quartile Range); unit: units on a scale] — mYPAS is an observational measure of children's preoperative anxiety consisting of 27 items divided into 5 categories: Activity, Vocalizations, Emotional Expressivity, State of Arousal and Use of Parent. Scores range from 22.5 to 100 with higher scores indicating greater anxiety.
  units on a scale | 28.3 [23.3 to 28.3] | 28.3 [23.3 to 28.3] | 28.3 [23.3 to 28.3]
Parental State-Trait Anxiety Inventory in preop [Median (Inter-Quartile Range); unit: units on a scale] — State-Trait Anxiety Inventory: Self-reported anxiety instrument containing two separate 2-item subscales that measure trait (baseline) and state (situational) anxiety. Range 20 to 80 with higher scores indicating greater anxiety.
  units on a scale | 36.0 [26.5 to 42.8] | 38.0 [31.0 to 45.0] | 36.0 [28.0 to 44.5]

OUTCOME MEASURES:

1. Primary Outcome: Perioperative Pediatric Anxiety (Change From Baseline)
Description: Modified Yale Preoperative Anxiety Scale (Observational measure of anxiety in five categories (activity, emotional expressivity, state of arousal, vocalization, and use of parents); Total range 0 to 100 with higher scores indicating greater anxiety)
Time Frame: (Day 0 + 15 minutes on average from initial baseline) On entering the OR
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 33 | 37
units on a scale | 0.0 [0.0 to 0.0] | 5.0 [0.0 to 10.0]

2. Primary Outcome: Perioperative Pediatric Anxiety (Change From Baseline)
Description: as for outcome 1
Time Frame: (Day 0 + 30 minutes on average from initial baseline) During mask induction
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 33 | 37
units on a scale | 0.0 [0.0 to 0.0] | 13.3 [5.0 to 26.7]

3. Secondary Outcome: Perioperative Parental Anxiety (Change From Baseline)
Description: State-Trait Anxiety Inventory: Self-reported anxiety instrument containing two separate 2-item subscales that measure trait (baseline) and state (situational) anxiety. Total range 20 to 80 with higher scores indicating greater anxiety. The value is a sum of trait and state anxiety.
Time Frame: (Day 0 + 45 minutes on average from initial baseline) After mask induction
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 33 | 37
units on a scale | 0 [-3 to 3] | 0 [-3 to 3]

4. Secondary Outcome: Induction Compliance Checklist
Description: Induction Compliance Checklist (An observational scale used to describe the compliance of a child during induction of anesthesia, range 0 to 11 with higher scores indicating less compliance)
Time Frame: (Day 0 + 30 minutes on average from initial baseline) During mask induction
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 33 | 37
units on a scale | 0 [0 to 0] | 0 [0 to 1]

5. Secondary Outcome: Parental Satisfaction
Description: 21-item parental satisfaction questionnaire after induction of general anesthesia (T3). Parental satisfaction score range: 21-84. Higher scores represent higher satisfaction.
Time Frame: (Day 0 + 45 minutes on average from initial baseline) After mask induction
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 33 | 37
units on a scale | 83 [76 to 84] | 80 [76 to 83]

6. Other Pre Specified Outcome: Anesthesia Length
Description: Length of time that patient received anesthesia care.
Time Frame: (Day 0 + 120 minutes on average from initial baseline) After exiting the OR
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 34 | 37
minutes | 80 (91) | 101 (119)

7. Other Pre Specified Outcome: Surgery Length
Description: Length of surgery from procedure start to procedure finish
Time Frame: (Day 0 + 120 minutes on average from initial baseline) After exiting the OR
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 34 | 37
Minutes | 62 (85) | 77 (106)

8. Other Pre Specified Outcome: Pre-medication Given
Description: Whether patient was given anxiolytic medication prior to induction of general anesthesia
Time Frame: (Day 0 + 30 minutes on average from initial baseline) On induction of anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 34 | 37
Participants
  Yes | 0 | 0
  No | 34 | 37

9. Other Pre Specified Outcome: Parent Present for Induction
Description: Whether parent was present in operating room during induction of anesthesia
Time Frame: (Day 0 + 30 minutes on average from initial baseline) On induction of anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Perioperative Virtual Reality Headset | Control
Number analyzed (Participants) | 34 | 37
Participants
  Yes | 30 | 35
  No | 4 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the perioperative period, generally ranging 2-4 hours after intervention or routine anesthetic induction.
Arm/Group | Perioperative Virtual Reality Headset | Control
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/37
Other Adverse Events (participants affected / at risk) | 0/33 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03583450/Prot_SAP_000.pdf